CLINICAL TRIAL: NCT01933412
Title: Efficacy and Safety of Sci B Vac vs. Engerix in Dialysis Patients
Brief Title: Efficacy and Safety of Hepatitis B Vaccine in Chronic Kidney Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Director of Institutional Research, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TLVMC1.2013
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Kidney Disease; Hepatitis B
Keywords: Dialysis; Hepatitis B
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sci-B-Vac Hepatitis B Vaccine (Experimental): Sci-B-Vac Hepatitis B Vaccine
  Interventions: Biological: Sci-B-Vac Hepatitis B Vaccine
- Engerix B Hepatitis B Vaccine (Active Comparator): Engerix B Hepatitis B Vaccine
  Interventions: Biological: Engerix B Hepatitis B Vaccine

INTERVENTIONS:
Biological: Sci-B-Vac Hepatitis B Vaccine — Sci-B-Vac Hepatitis B Vaccine
  Arms: Sci-B-Vac Hepatitis B Vaccine
Biological: Engerix B Hepatitis B Vaccine
  Arms: Engerix B Hepatitis B Vaccine

SUMMARY:
This is an open label clinical study designed to evaluate the safety and immunogenicity of Sci-B-Vac Hepatitis B Vaccine compared to Engerix-B Hepatitis B Vaccine in dialysis patients. The study hypothesis is that vaccination with Sci B Vac will achieve a higher seroprotection rate and a higher anti-Hepatitis B surface antibody serum titer level than vaccination with Engerix-B Dialysis patients will be categorized as "naïve" or "previously vaccinated" and each group will be randomized to treatment. Naïve patients randomized to Sci-B-Vac Hepatitis B vaccine will receive vaccination in three doses, 10 μg each, at 0, 1, and 6 months, or Engerix-B Hepatitis B vaccine given in four doses, 40 μg each, at 0, 1, 2, and 6 months. Previously vaccinated patients randomized to Sci-B-Vac Hepatitis B vaccine will receive vaccination in three doses, 20 μg each, at 0, 1, and 6 months, or Engerix-B Hepatitis B vaccine given in four doses, 40 μg each, at 0, 1, 2, and 6 months. All vaccines will be administered via intra-muscular injection to the deltoid muscle. The study will consist of three periods: a screening period of up to four weeks, a 24-week open-label treatment period, and a 24-week safety follow-up period. The total expected duration of the study per subject is 52 weeks as follows: Screening period: approximately 4 weeks; treatment period: 24 weeks; and follow up period: 24 weeks. The primary endpoint is the by-vaccine difference in the proportion of subjects attaining seroprotective immune response (anti-Hepatitis B surface antibody ≥ 10 IU/mL) 4 weeks after the last vaccination with either Sci-B-Vac or Engerix-B. Secondary endpoints include anti-Hepatitis B surface antibody geometric mean concentrations calculated for all subjects upon last active dose; the proportion of subjects with anti-Hepatitis B surface antibody concentrations equal to or above 10 IU/mL for all subjects at 12 weeks following the first vaccine dose; the by-treatment difference in serum titer levels of anti-Hepatitis B surface antibodies at 12, 24 and 52 weeks following the first vaccination. A by-vaccine comparison of adverse events will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Three months dialysis treatment for Chronic Kidney Disease; anti-Hepatitis B surface antibody titer levels < 10 IU/ml

Exclusion Criteria:

* anti-Hepatitis B surface antibody titer levels > 10 IU/ml
* Hepatitis B surface antigen positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
anti-Hepatitis B surface levels ≥ 10 IU/mL | 28 weeks
  The by-vaccine difference in the proportion of subjects attaining seroprotective immune response (anti-Hepatitis B surface antibody ≥ 10 IU/mL) 4 weeks after the last vaccination with either Sci-B-Vac or Engerix-B.

SECONDARY OUTCOMES:
anti-Hepatitis B surface antibody Geometric Mean Concentrations | 24 weeks
  By vaccine comparison of anti-Hepatitis B surface antibody Geometric Mean Concentrations calculated for all subjects upon last active dose
52 week anti-Hepatitis B surface antibody Geometric Mean Concentrations | 52 weeks
  By-vaccine comparison of anti-Hepatitis B surface antibody Geometric Mean Concentrations calculated for all subjects at week 52
serum titer levels of anti-Hepatitis B surface antibodies | 12, 24 and 52 weeks
  The by-treatment difference in serum titer levels of anti-Hepatitis B surface antibodies at 12, 24 and 52 weeks following the first vaccination.
Adverse events | 12, 24 and 52 weeks
  Spontaneous and elicited reports of all adverse events in all body systems.

CONTACTS AND LOCATIONS:
Overall Officials: Talia Weinstein, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center Dialysis Unit, Tel Aviv, Israel